CLINICAL TRIAL: NCT06101875
Title: Feasibility of Targeted Health Coaching for Patients With Low Activation Waiting for Total Hip or Total Knee Replacements
Brief Title: Health Coaching for Patients Waiting for Hip or Knee Replacements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ER53641774
Record Dates: First submitted 2023-09-29; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Hip; Osteo Arthritis Knee
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching (Experimental): Patients will be assigned a health coach and be eligible to 8 sessions over a 12 week period.
  Interventions: Other: Health Coach (Health coaching)
- Control (Active Comparator): Patients will be enrolled onto the digital toolkit.
  Interventions: Other: Digital Toolkit (Control)

INTERVENTIONS:
Other: Health Coach (Health coaching) — Patients will be assigned a health coach and be eligible to 8 times, 1 hour sessions over a 12 week period. The health coach will use techniques to increase their ability to self-manage, motivation levels and commitment to change their behaviour.
  Arms: Health Coaching
Other: Digital Toolkit (Control) — This is an online website, unsupervised, 12-week self-management programme.
  Arms: Control

SUMMARY:
A randomised controlled feasibility study of a health coaching intervention targeting people on the waitlist for hip or knee replacement surgery with low patient activation.

DETAILED DESCRIPTION:
Determine the feasibility of recruitment and retention to the trial. Evaluate the acceptability of research procedures and outcome measures. Explore the impact of trial participation through patient activation, self-reported health outcomes and interviews.

ELIGIBILITY:
Inclusion Criteria:

* On the waitlist for total hip or total knee replacement surgery
* PAM level 1 or 2

Exclusion Criteria:

* Current participation in care with a focus on self-management education
* PAM Level 3 or 4

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-11-14 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rates | 4 weeks
  Defined as rate of invited participants who are eligible and consenting.
Retention Rates | 12 weeks
  Retention rates will be established as discontinuation with the exercise intervention and absence from the assessment sessions.
Acceptability of intervention | 12 weeks
  Will be evaluated by participants feedback via one-to-one semi-structured interviews.
Competition rates | 12 weeks
  Completion is determined by participants that attend baseline and follow-up testing.

SECONDARY OUTCOMES:
Change in patient activation | 12 weeks
  Patient activation measure 13-item questionnaire (0 - 100 point scale)
Change in quality of life | 12 weeks
  EQ-5D-5L questionnaire (1 - 5 point scale)
Change in pain score | 12 weeks
  Oxford score questionnaire (0 - 48 point scale)
Change in physical activity | 12 weeks
  IPAQ-SF questionnaire (MET/mins)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Maden-Wilkinson, PhD, Principal Investigator — Sheffield Hallam Unviersity
Locations (1):
- Sheffield Hallam University, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No